CLINICAL TRIAL: NCT00588341
Title: Phase II Trial of Neoadjuvant Temozolomide in Melanoma Patients With Palpable Stage III or IV Disease Undergoing Complete Surgical Resection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-076
Record Dates: First submitted 2007-12-26; First posted 2008-01-08 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2015-12

CONDITIONS: Melanoma; Skin Cancer; Cancer
Keywords: Melanoma; Skin Cancer; Cancer; Temozolamide; TMZ
MeSH Terms: conditions — Melanoma; Skin Neoplasms; Neoplasms | interventions — Temozolomide

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — At the start of the trial a core needle biopsy of a palpable tumor will be obtained percutaneously in the office after administration of local anesthesia. Patients will then be treated with TMZ according to the extended dosing schedule of 75mg/m2/day x 6 weeks every 8 weeks. After each cycle, patients will be re-evaluated for response.
  Responding patients will be offered another cycle of treatment. Patients will be treated until best response, progression of disease, or 6 cycles, whichever comes first.
  After completing temozolomide treatment, patients will be evaluated for surgical resection. It is expected that, unless there is progression of disease, patients will undergo resection (i.e. therapeutic lymph node dissection). In patients who have a complete clinical response to temozolomide, whether or not to do a subsequent lymph node dissection will be left up to the discretion of the surgeon and the patient.
  Other Names: TMZ

SUMMARY:
In this study, we want to find out how likely it is for temozolomide to shrink melanoma tumors that have spread only to areas that could be removed by surgery. We also want to study the melanoma before and after temozolomide treatment to learn why some tumors respond and others do not. This is a Phase II trial. This means that it will test a drug - in this case, temozolomide -- that has already been studied and shown to be safe.

Surgery, when possible, is the main treatment for patients with melanoma like yours. In most people, however, melanoma cells have already spread to other places in the body. This means that even with surgery, many people will have the melanoma come back. This is often fatal.

One goal of this trial is to treat the melanoma cells that might have spread before they have a chance to grow.

As part of this trial, we also study which genes are turned on and which genes are turned off in your tumor. We will obtain tumor from the biopsy done before you started temozolomide treatment and from the tumor removed during the surgery done after you finish temozolomide treatment. This may help us understand how temozolomide works and how to recognize which tumors will respond.

Before and during the temozolomide treatment, we will also test a new way of measuring the amount of tumor present. This involves a special way of analyzing the CT scan which you will have anyway. This new technique may allow us to see tumor shrinkage very early in the treatment course.

DETAILED DESCRIPTION:
In this Phase II trial, chemotherapy-naïve patients with palpable Stage III or Stage IV M1a melanoma scheduled to undergo surgical resection will be treated with TMZ in 8 week cycles according to the extended dosing schedule of 75mg/m2/day x 6 weeks with 2 weeks off. Patients will be treated until maximal response to TMZ and then undergo resection of residual disease. The primary endpoint will be tumor response as measured by the RECIST criteria. Patients will be seen monthly.

ELIGIBILITY:
Inclusion Criteria:

* Palpable Stage III (N1b, N2b, N2c, or N3) or Stage IV (M1a) cutaneous melanoma. Patient must be a potential candidate for complete surgical resection.
* Age ≥ 18 years
* Histologic proof of pathology reviewed and confirmed at MSKCC
* Measurable disease by RECIST criteria
* Determination of surgical resectability by surgeon at MSKCC
* No prior chemotherapy for melanoma. Prior interferon, interleukin-2 or vaccine therapy is allowed.
* No other concurrent chemotherapy, immunotherapy, or radiotherapy
* Karnofsky performance status ≥60
* Adequate organ function

Exclusion Criteria:

* Uveal or mucosal melanoma
* Patients with melanoma deemed not amenable to surgical resection or who are not surgical candidates for medical reasons
* Frequent vomiting or medical conditions that could interfere with oral medication intake
* Serious infection requiring antibiotics, or nonmalignant medical illnesses that are uncontrolled or whose control might be jeopardized by the complications of this therapy
* Pregnancy or nursing
* History of HIV infection even if on HAART as TMZ leads to CD4+ T cell leukopenia
* Concurrent use of high dose vitamins and herbs
* Other on-going investigational therapy, concurrent chemotherapy, immunotherapy or radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Chapman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering web site — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Temozolomide: Patients will then be treated with TMZ according to the extended dosing schedule of 75mg/m2/day x 6 weeks every 8 weeks.
Period: Overall Study
Arm/Group | Treatment
Started | 24
Completed | 19
Not Completed | 5
Not completed — Withdrawal by Subject | 3
Not completed — Not treated due to metastatic disease | 1
Not completed — Patient ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response (Complete Response or Partial Response)
Description: The Response Evaluation Criteria in Solid Tumors (RECIST) will be used to determine treatment response.
  Clinical Complete Response (CRc) Disappearance of all target lesions and non-measurable disease.
  Pathological Complete Response (CRp) A CRc in which a lymph node dissection done after completing temozolomide treatment shows no pathological evidence of melanoma. Partial Response (PR) A greater or equal then 30% in the sum of the longest diameter of all target lesions relative to baseline measurement
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 19
participants
  Complete Response (CR) | 2
  Partial Response (PR) | 2
  Non Responder | 15

ADVERSE EVENTS:
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 22/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=24)
Fatigue (General disorders) | 22 (22)
Nausea (Gastrointestinal disorders) | 22 (22)
Vomiting (Gastrointestinal disorders) | 22 (22)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes